CLINICAL TRIAL: NCT02905734
Title: Nicotine Replacement Therapy in Nicotine-dependent Arrestees: a Monocentric Randomized Simple Blind Study
Brief Title: Nicotine Replacement Therapy in Nicotine-dependent Arrestees
Acronym: SUBNIGAV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P 140703
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Nicotine Dependence
Keywords: Nicotine replacement therapy; Tobacco
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nicotine replacement patch (Experimental): Single administration of a nicotine patch (14 mg or 21 mg, according to the Heaviness of Smoking Index)
  Interventions: Drug: Nicotine patch
- placebo patch (Placebo Comparator): Single administration of a placebo patch
  Interventions: Other: placebo patch

INTERVENTIONS:
Drug: Nicotine patch — Single administration of an active treatment (nicotine patch)
  Other Names: NICOPATCH; NICOPATCHLIB
  Arms: nicotine replacement patch
Other: placebo patch — Single administration of a placebo treatment
  Other Names: duoderm spot; TEGADERM
  Arms: placebo patch

SUMMARY:
Tobacco use affects more than 50% of adult arrestees, of which 70% are dependent on nicotine. However, they have no access to tobacco during detention in police cells. Nicotine withdrawal symptoms, that include irritability, anxiety and lack of concentration, may worsen the arrestee's health status during detention. Nicotine withdrawal is a treatable condition. Validated treatments in other situations than police custody include nicotine replacement therapy.

This study is based on the following hypotheses: Manifestations related to nicotine withdrawal could increase the discomfort due to detention in police cells, A nicotine replacement therapy initiated during detention could improve the course of detention in police cells and could be useful in a perspective of long-lasting smoking cessation.

The primary objective is to evaluate the efficacy of nicotine replacement therapy among nicotine-dependent arrestees on the course of detention as perceived by the arrestees. Our secondary objectives are to evaluate the efficacy of nicotine replacement therapy on desire to smoke during detention in police cells and to improve long-term smoking cessation among dependent smokers.

Interventions consist in the single administration of an active treatment (nicotine patch) or of a control treatment (placebo patch). Evaluations will include the results of a medical examination during detention, a self evaluation by the arrestees of their desire to smoke, and medical consultations and evaluations of tobacco use 7-10 days, one month and six months later.

DETAILED DESCRIPTION:
Police custody is a matter of significant public attention in France, as approximately 700,000 people are detained in police cells each year in this country.

Tobacco use affects more than 50% of adult arrestees, of which 70% are dependent on nicotine. However, they have no access to tobacco during detention in police cells. Nicotine withdrawal symptoms, including irritability, anxiety and lack of concentration, may worsen the arrestee's health status during detention. Nicotine withdrawal is a treatable condition. Validated treatments in other situations than police custody include nicotine replacement therapy. Available medical guidelines in police custody do not mention nicotine dependence.

This study is based on the following hypotheses: (1) Manifestations related to nicotine withdrawal could increase discomfort due to the detention in police cells, (2) A nicotine replacement therapy initiated during detention could improve the course of detention in police cells and (3) could be useful in a perspective of long-lasting smoking cessation.

The primary objective is to evaluate the efficacy of nicotine replacement therapy among nicotine-dependent arrestees on the course of detention as perceived by the arrestees. The secondary objectives are to evaluate the efficacy of nicotine replacement therapy on desire to smoke during detention in police cells and to improve long-term smoking cessation among dependent smokers.

Interventions consist in the single administration of an active treatment (nicotine patch) or of a control treatment (placebo patch). Evaluations will include the results of a medical examination during detention, a self-assessment by the arrestees of their desire to smoke, and medical consultations and evaluations of tobacco use 7-10 days, one month and six months later.

Primary endpoint: self-assessment of detention course by the arrestee (Likert scale).

Secondary endpoints: Desire to smoke during detention in police cells (Likert scale); willingness to change their tobacco use (Likert scale); tobacco use at 1 and 6 months.

Methods:

The study design includes two parts. The first part will be the intervention (patch administration) during detention in police cells: single blind randomized administration of a nicotine patch or a placebo patch. The second part will be observational and include follow-up evaluations at 7-10 days, 1 month and 6 months.

The active treatment will consist of a single administration of nicotine patches (21 mg/24h or 14 mg/24h according to the Heaviness of smoking index [HIS], 21 mg for those with HSI>3, 14 mg for those with HSI of 1 or 2). The control treatment will be a non-active placebo patch.

Number of participants: 1000 (two groups of 500). The total duration of the study will be 33 months.

ELIGIBILITY:
Inclusion Criteria:

* Arrestees examined by a physician during detention in police cells
* aged 18 or older
* smoking at least 10 cigarettes per day
* giving written consent to participate in the study
* health status compatible with detention in police cells

Exclusion Criteria:

* Lack of understanding of the study
* contra-indication to nicotine replacement therapy
* health status incompatible with detention in police cells
* serious mental disorder
* usual place of residence outside Seine-Saint-Denis

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Perceived quality of detention in police cells at 8 hours following treatment administration | 8 hours maximum after treatment
  self-assessment of detention course by the arrestee (Likert scale).

SECONDARY OUTCOMES:
Rating of desire to smoke after treatment administration | 8 hours maximum after treatment
  Desire to smoke during detention in police cells (Likert scale)
Rating of intention to quit smoking after treatment administration; | 8 hours maximum after treatment
  willingness to change their tobacco use (Likert scale)
Mean number of cigarettes per day at one month | one month after treatment
  tobacco use at 1 month consultation
Mean number of cigarettes per day at six months | six months after treatment
  tobacco use at 6 months consultation

CONTACTS AND LOCATIONS:
Overall Officials: Patrick CHARIOT, MD, Principal Investigator — Hospital Jean Verdier
Locations (1):
- Médecine légale - Hôpital Jean Verdier, Bondy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chariot P, Lepresle A, Lefevre T, Boraud C, Barthes A, Tedlaouti M. Alcohol and substance screening and brief intervention for detainees kept in police custody. A feasibility study. Drug Alcohol Depend. 2014 Jan 1;134:235-241. doi: 10.1016/j.drugalcdep.2013.10.006. Epub 2013 Oct 23. PMID 24210771
- [Background] Chariot P, Beaufrere A, Denis C, Dang C, Vincent R, Boraud C. Detainees in police custody in the Paris, France area: medical data and high-risk situations (a prospective study over 1 year). Int J Legal Med. 2014 Sep;128(5):853-60. doi: 10.1007/s00414-014-0990-4. Epub 2014 Mar 27. PMID 24671410
- [Background] Cropsey KL, Jones-Whaley S, Jackson DO, Hale GJ. Smoking characteristics of community corrections clients. Nicotine Tob Res. 2010 Jan;12(1):53-8. doi: 10.1093/ntr/ntp172. Epub 2009 Dec 8. PMID 19996145
- [Background] Richmond R, Indig D, Butler T, Wilhelm K, Archer V, Wodak A. A randomized controlled trial of a smoking cessation intervention conducted among prisoners. Addiction. 2013 May;108(5):966-74. doi: 10.1111/add.12084. Epub 2013 Mar 11. PMID 23228222
- [Background] Tzelepis F, Paul CL, Walsh RA, Knight J, Wiggers J. Who enrolled in a randomized controlled trial of quitline support? Comparison of participants versus nonparticipants. Nicotine Tob Res. 2013 Dec;15(12):2107-13. doi: 10.1093/ntr/ntt114. Epub 2013 Aug 3. PMID 23911847